CLINICAL TRIAL: NCT02541214
Title: Evaluation of a Nasal Mask for the Treatment of Obstructive Sleep Apnea in New Zealand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-171
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Trial Nasal Mask (Experimental): The participant will use the Saturn nasal mask for 2 weeks in home
  Interventions: Device: Trial Nasal Mask

INTERVENTIONS:
Device: Trial Nasal Mask

SUMMARY:
Currently, Fisher and Paykel Healthcare (FPH) is developing a new nasal mask.

This investigation is designed to evaluate the performance of the trial nasal mask, focused specifically on how the different seal sizes will perform on Obstructive Sleep Apnea participants who are currently on Positive Airway Pressure therapy.

Participant's prescribed treatment pressure with their usual mask will be collected for 7 days ± 3 days prior to mask fitting with the trial nasal mask. They will then be issued with the trial nasal mask to use in-home for 14 days ± 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Diagnosed with Ostructive Sleep Apnea by a practicing physician or clinicans
* Existing nasal or nasal pillows user
* Prescribed Positive Airway Pressure therapy (Bi-Level or Continuous Positive Airway Pressure (CPAP) or Automatic Positive Airway Pressure (APAP))

Exclusion Criteria:

* Inability to give informed consent
* Pregnant or think they may be pregnant
* Anatomical or physiological conditions making Positive Airway Pressure therapy inappropriate (e.g unconsolidated facial fracture)
* Patients who are in a coma or decreased level of consciousness
* Current diagnosis of CO2 retention
* Commercial Drivers who are investigated by New Zealand Transport Agency (NZTA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Subjective measurements of comfort on the trial Nasal Mask gathered through a custom questionnaire | 2 weeks in home

SECONDARY OUTCOMES:
Seal performance of the trial Nasal mask as measured by the subjective perception of leak through a custom questionnaire, in addition to objective leak data and treatment efficacy through the Positive Airway Pressure therapy device. | 2 weeks in home
  the participant would choose from a 5 point likert scale on a questionnaire. The scale range from "very good" to "very poor"
Objective leak data through the Positive Airway Pressure therapy device | 2 weeks in home
  Evaluating the leak of the trial Nasal mask
Treatment efficacy through the Positive Airway Pressure therapy device | 2 weeks in home
  Evaluating the number of apnea/hypopnea per hour
Preference of the Trial Nasal mask compared to the participant's usual mask through a custom questionnaire. | 2 weeks in home
  the participant would either choose the trial Nasal mask or their usual mask as their primary mask

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Waikato District Health Board, Hamilton
  - Hawke's Bay District Health Board, Hastings